CLINICAL TRIAL: NCT00002294
Title: Double Blind Placebo Controlled Study of Fluconazole (UK-49,858) for Maintenance Treatment of Cryptococcal Meningitis in Patients With Acquired Immunodeficiency Syndrome
Brief Title: A Study of Fluconazole in the Treatment of Cryptococcal Meningitis in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 012A; 056-114A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-12

CONDITIONS: Meningitis, Cryptococcal; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Fluconazole; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections; AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Acquired Immunodeficiency Syndrome | interventions — Fluconazole

INTERVENTIONS:
Drug: Fluconazole

SUMMARY:
To compare the safety and effectiveness of fluconazole with that of placebo as maintenance treatment for preventing the relapse of cryptococcal meningitis in patients with AIDS.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiviral therapy (e.g., zidovudine).
* Prophylaxis (including aerosolized pentamidine) for Pneumocystis carinii pneumonia (PCP).

Concurrent Treatment:

Allowed:

* Radiation therapy for mucocutaneous Kaposi's sarcoma.

Patients must be oriented to person, place, and time and able to give written informed consent.

* Patients must have had an acute episode of cryptococcal meningitis that was documented by recovery and identification of cryptococcus from lumbar cerebrospinal fluid (CSF) culture within 4 months of study entry.
* Adequate therapy will consist of 6 - 16 weeks of treatment with amphotericin B alone, amphotericin B + oral flucytosine, or a period of the combination followed by amphotericin alone. Adequate regimens will include:
* A minimum total amphotericin B dose of 2 grams as monotherapy.
* 6 weeks of flucytosine at 150 mg/kg/day (or levels of 20 to 100 mcg/ml demonstrated) plus amphotericin B at an average daily dose of at least 0.3 mg/kg/day or to a total dose of 1 gram.
* After a shorter period of the combination amphotericin/flucytosine therapy, an additional Y grams of amphotericin B monotherapy will make therapy adequate where Y = 2 gm-(X weeks combination therapy / 3 weeks).
* For example, a patient who received 3 weeks of combination followed by amphotericin alone would need an additional 2 gm - 3 weeks/3 weeks = 1 gm of amphotericin B.
* Patients need not be receiving amphotericin B at the time of randomization but must begin study maintenance therapy within 3 weeks of cessation of primary amphotericin B therapy.

Prior Medication:

Allowed:

* Antiviral therapy (e.g., zidovudine (AZT)).
* Prophylaxis (including aerosolized pentamidine) for Pneumocystis carinii pneumonia (PCP).

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Clinical evidence of acute or chronic meningitis based upon any etiology other than cryptococcosis.
* History of allergy or intolerance of imidazoles, azoles, or amphotericin B.
* Moderate or severe liver disease.

Concurrent Medication:

Excluded:

* Intrathecal amphotericin B.
* Coumarin-type anticoagulants.
* Oral hypoglycemics.
* Barbiturates.
* Phenytoin.
* Immunostimulants.
* Investigational drugs or approved (licensed) drugs for investigational indications.

Concurrent Treatment:

Excluded:

* Lymphocyte replacement.

Patients with the following are excluded:

* Clinical evidence of acute or chronic meningitis based upon any etiology other than cryptococcosis.
* History of allergy or intolerance of imidazoles, azoles, or amphotericin B.
* Moderate or severe liver disease defined by specific lab values.
* Inability to take oral medications reliably.

Prior Medication:

Excluded:

* Intrathecal amphotericin B.
* Coumarin-type anticoagulants.
* Oral hypoglycemics.
* Barbiturates.
* Phenytoin.
* Immunostimulants.
* Investigational drugs or approved (licensed) drugs for investigational indications.

Prior Treatment:

Excluded:

* Lymphocyte replacement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Dr Robert Larsen, Los Angeles, California
  - UCI Med Ctr, Orange, California
  - UCSD, San Diego, California
  - Dr Paul Rothman, Sherman Oaks, California
  - Stanford Univ School of Medicine, Stanford, California